CLINICAL TRIAL: NCT02501642
Title: Smart Phone Application for Postconcussion Symptom Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 13-196
Record Dates: First submitted 2015-07-02; First posted 2015-07-17 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concussion Coach group (Experimental): After informed consent and randomization, participants will complete baseline study measures and will receive an iPod touch® with the Concussion Coach "Explorer" version
  Interventions: Behavioral: Concussion Coach
- Treatment as usual (Other): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Concussion Coach — smart phone app with educational material on postconcussion symptoms and behavioral self-monitoring/strategies
  Arms: Concussion Coach group
Other: Treatment as usual — Treatment as usual
  Arms: Treatment as usual

SUMMARY:
The proposed study will address a very important issue for the VA both currently and in the future -- the high percentage of OIF/OEF/OND Veterans who have been medically diagnosed with a mild traumatic brain injury (mild TBI) and experience distressing symptoms. "Smart phone" mobile applications have become a primary source of information and communication among large percentages of Americans, especially those of the OIF/OEF/OND generation. The proposed study is a 4-year randomized control trial investigating the utility of an interactive, self-management smartphone application, "TBI Coach," one of a suite of mobile applications developed by VA. The primary goal of the proposed study is to evaluate the efficacy of TBI Coach for improving clinical outcomes in those with a history of mild TBI and to determine what aspects of TBI Coach are most useful to Veterans. An overarching goal of this line of research is to improve access among Veterans with mild TBI who still have symptoms months to years after injury.

Objectives. The study will pursue the following objectives:

1. Evaluate the efficacy of TBI coach for improving clinical outcomes among recipients of TBI Coach.
2. Determine the aspects of TBI Coach most associated with positive outcomes.
3. Obtain qualitative information on factors associated with use of TBI coach or with deriving benefit from use of TBI Coach that can be used to inform future modifications of the application and wide scale implementation.

DETAILED DESCRIPTION:
Patients who meet eligibility criteria and consent to participate in the study will be randomly assigned to one of two arms, either the Concussion Coach group, which will receive an iPod touch® with the Concussion Coach "Explorer" version, or into the no mobile app control group. Study personnel will explain the purpose of the study, complete the informed consent process, obtain the random treatment assignment from a randomization sheet, and introduce the participant to his/her baseline evaluator. The random assignment to intervention will be accomplished in blocks within each site. While small block sizes allow intervention group sizes to be very similar it may make the allocation process predictable. Therefore to reduce selection bias and achieve balance across the intervention arms sequence list of individual assignments by random block sizes will be generated.

Both groups will be assessed in a pre/post intervention design and will be compensated for their time completing study surveys. During the 3 months that they are involved in the study, the intervention group will be sent (via Concussion Coach) reminders to engage with the app on a weekly basis. Their use (e.g., total time spent on each component of the app) will be collected electronically. Both groups will receive care as usual (meaning their regularly scheduled VA appointments and medications). At the completion of the study, both groups will be encouraged to download the App for their own use, with assistance from the study team if needed.

Description of Intervention & Training The Concussion Coach is designed to provide psychoeducation, self-assessment, and treatment of PCS symptoms following a mild TBI. The PI and three of the co-investigators were co-developers of Concussion Coach. The public-facing Concussion Coach will be available for free download from a public marketplace and available for use with most mobile devices. The application has the advantage of privacy and anonymity, thus addressing the stigma often expressed as a barrier to seeking treatment. A mirror version of the public version, called Concussion Coach "Explorer Version", will be developed within three months and used for this study. Unlike the public version, it will have the capacity to collect usage information, such as length of time spent on each part of the app, self-report ratings of symptoms and distress, and identification of "favorites" among the self-help tools. These data can be uploaded in a de-identified form to a HIPAA compliant server. Other than the ability to collect data, it will be exactly like the "real" Concussion Coach. The Explorer version will be developed by our collaborators, Vertical Product Development, which developed Concussion Coach, PTSD Coach, and PTSD Explorer version. Explorer versions are especially useful as they allow for unobtrusive, highly detailed, real-time data collection without relying on patient self-report. In addition, the Concussion Coach will be an 'opportunistic' exporter of data. It will upload data to the server whenever it has new data and is in a WiFi zone; participants do not have to have a home wireless network. If they never enter a WiFi area, the investigators will collect their data at study termination when the investigators collect the iPod touch®. The investigators will utilize ohmage, an existing open source technology stack, to port the app to the server.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* History of mild TBI (DoD/VA) as determined by trained, experienced staff via interview and medical record review via comprehensive evaluation process within PNS with current symptoms complaints operationally defined as at least two symptoms on the NSI endorsed at the 'moderate' level or a total score on the NSI greater than 25
* Must speak and read English
* Not have a history of moderate to severe TBI
* Not have a self-reported diagnosis of psychosis or be actively suicidal

Exclusion Criteria:

* Subjects who report prior experience with Concussion Coach will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy S Kretzmer, PhD BA, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (2):
- United States (2):
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
To allow collaboration of information with other interested parties who may be researching the use of Apps for TBI Veterans.

REFERENCES:
- [Result] Bradley SE, Haun J, Powell-Cope G, Haire S, Belanger HG. Qualitative assessment of the use of a smart phone application to manage post-concussion symptoms in Veterans with traumatic brain injury. Brain Inj. 2020 Jul 2;34(8):1031-1038. doi: 10.1080/02699052.2020.1771770. Epub 2020 Jun 4. PMID 32493066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment closed on 9.30.2018
Pre-assignment Details: Enrollment closed on 9.30.2018 N/A
Period: Overall Study
Arm/Group | Concussion Coach Group | Treatment as Usual
Started | 238 (Start of study: 10.1.2014) | 241 (Start of study: 10.1.2014)
Completed | 231 (Study ended 9.30.2018) | 230 (Study ended 9.30.2018)
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concussion Coach Group | Treatment as Usual | Total
Number analyzed (Participants) | 238 | 241 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 238 | 241 | 479
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (16) | 35 (15) | 35.5 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: missing data for gender
  Participants
    number analyzed (Participants) | 230 | 228 | 458
    Female | 21 | 21 | 42
    Male | 209 | 207 | 416
Race (NIH/OMB) [Count of Participants; unit: Participants] — Enrollment ended 9.30.2018
  Participants
    American Indian or Alaska Native | 2 | 1 | 3
    Asian | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 2 | 13 | 15
    Black or African American | 37 | 41 | 78
    White | 183 | 171 | 354
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 10 | 13 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 238 | 241 | 479

OUTCOME MEASURES:

1. Primary Outcome: Neurobehavioral Symptom Inventory
Description: The Neurobehavioral Symptom Inventory is a 22-item questionnaire developed to evaluate post-concussive symptom severity following mild TBI (Cicerone and Kalmar 1995). Participants are asked to rate each symptom on a scale of 0-4 (None, Mild, Moderate, Severe, Very Severe) with three different categories of symptoms: Affective/psychological/stress, somatic/physical and cognitive (reflecting three factors). Scores can range from 0-88, with higher scores indicating more severe symptom endorsement.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Concussion Coach Group | Treatment as Usual
Number analyzed (Participants) | 231 | 230
score on a scale | 33 (16) | 33 (17)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout study collection period, 36 months.
Arm/Group | Concussion Coach Group | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/238 | 0/241
Serious Adverse Events (participants affected / at risk) | 0/238 | 0/241
Other Adverse Events (participants affected / at risk) | 0/238 | 0/241

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT02501642/Prot_SAP_000.pdf